CLINICAL TRIAL: NCT02611674
Title: Methodology Study of Novel Electrophysiological, Physical, and Imaging Outcome Measures to Assess the Progression of Amyotrophic Lateral Sclerosis
Brief Title: Methodology Study of Novel Outcome Measures to Assess Progression of ALS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 999AS003
Record Dates: First submitted 2015-10-08; First posted 2015-11-23 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of the study are to estimate and rank-order the longitudinal standardized mean changes over 6 months and over 12 months, for a set of outcome measures administered to participants with amyotrophic lateral sclerosis (ALS), in order to identify measures that are more sensitive to disease progression than Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R). The secondary objectives of this study are: To evaluate the test-retest reproducibility of each outcome measure; To determine correlations between 6 and 12-month changes in all exploratory measures with 18 and 24-month changes in ALSFRS-R and survival; To assess correlations between/among the various measures; To obtain biological samples in order to identify molecular correlates to the clinical measures and to further characterize previously identified and novel molecular biomarkers of disease progression for incorporation into future clinical studies.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of sporadic or familial ALS
* ALS onset within ≤5 years
* Must be 16 to 85 years of age, inclusive, for sites in the United States and 18 to 85 years of age, inclusive, for all sites outside of the United States

Key Exclusion Criteria:

* History of or positive test result at Screening for human immunodeficiency virus (HIV)
* History of or positive test result at Screening for hepatitis C virus (HCV) antibody or hepatitis B virus (HBV)
* Possibility of neuromuscular weakness other than ALS
* Unspecified reasons that, in the opinion of the site Investigator, make the subject unsuitable for enrollment or unlikely to be able to complete, at a minimum, the Month 6 Visit

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants suffering from ALS are recruited by participating physicians in a standard clinical practice setting.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal standardized mean change in electrophysiological measures as assessed by electrical impedance myography (EIM) | Baseline to Month 6 and Baseline to Month 12
  EIM is an electrophysiological technique in which current is applied to a muscle of interest and resultant voltage and impedance are measured. These measured parameters reflect the conductivity of underlying tissue and presumably the pathologic state of denervated muscle in an ALS participant
Longitudinal standardized mean change in electrophysiological measures as assessed by compound muscle action potential (CMAP) | Baseline to Month 6 and Baseline to Month 12
  CMAP is a standard electrophysiological measure generated by maximally stimulating a nerve such that all muscle fibers innervated by the respective nerve are depolarized. Reduction of CMAP amplitude reflects loss of motor axons and, therefore, is directly relevant to ALS.
Longitudinal standardized mean change in electrophysiological measures as assessed by motor unit number estimation (MUNE) | Baseline to Month 6 and Baseline to Month 12
  Optional, to be administered at each site's Investigator's discretion. MUNE is used to estimate the number of functioning motor units.
Longitudinal standardized mean change in electrophysiological measures as assessed by motor unit number index (MUNIX) | Baseline to Month 6 and Baseline to Month 12
  MUNIX estimates functioning motor units within a muscle. CMAP and surface electromyography potentials (surface interference patterns) are obtained at various levels of voluntary effort, and MUNIX is estimated using power and area of CMAP and surface interference patterns.
Longitudinal standardized mean change in muscle strength measures as assessed by hand-held dynamometry (HHD) | Baseline to Month 6 and Baseline to Month 12
  HHD tests isometric strength of multiple muscles using standard participant positioning. Approximately 10 muscle groups will be examined (per each side) in both upper and lower extremities.
Longitudinal standardized mean change in respiratory measures as assessed by slow vital capacity (SVC) | Baseline to Month 6 and Baseline to Month 12
  Vital capacity will be measured by means of an SVC test, administered in the upright position. Upright SVC will be determined by performing 3 to 5 measures, in accordance with criteria established by the American Thoracic Society and the European Respiratory Society.
Longitudinal standardized mean change in functional measures as assessed by Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | Baseline to Month 6 and Baseline to Month 12
  The ALSFRS-R has been demonstrated to predict survival. The ALSFRS-R measures 4 functional domains, including respiratory, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48 [Cedarbaum 1999], with higher scores representing better function.

SECONDARY OUTCOMES:
Within-participant test-retest reliability between the 2 repeated measurements occurring on Day 1 and Day 7 for EIM | Day 1 and Day 7
Within-participant test-retest reliability between the 2 repeated measurements for CMAP | Day 1 and Day 7
Within-participant test-retest reliability between the 2 repeated measurements for MUNE | Day 1 and Day 7
Within-participant test-retest reliability between the 2 repeated measurements for MUNIX | Day 1 and Day 7
Within-participant test-retest reliability between the 2 repeated measurements for HHD | Day 1 and Day 7
Within-participant test-retest reliability between the 2 repeated measurements for SVC | Day 1 and Day 7
Within-participant test-retest reliability between the 2 repeated measurements for ALSFRS-R | Day 1 and Day 7
Comparison between 6 and 12-month changes in exploratory measures with 18 and 24-month changes in ALSFRS-R and survival | Baseline to Month 24
Comparison between 6-month changes for muscle electrophysiological measures | Baseline to Month 12
Comparison between 6-month changes for muscle strength measures | Baseline to Month 12
Comparison between 6-month changes for functional measures | Baseline to Month 12
Comparison of molecular biomarkers with disease progression | Baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (21):
- United States (8):
  - University of California San Diego Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of South Florida, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, MA, Charlestown, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute Clinical Research Unit, Montreal, Quebec
- France (2):
  - Hopital Gui de Chauliac, Service de Neurologie, Montpellier, Hérault
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
- Germany (4):
  - Charite - Campus Virchow-Klinikum, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Ulm, Ulm
- Beaumont Hospital, Dublin, Ireland
- UMC Utrecht, Utrecht, CX, Netherlands
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- Royal Hallamshire Hospital, Sheffield, West Midlands, United Kingdom